CLINICAL TRIAL: NCT00296088
Title: A Prospective Observational Study of the Association Between Excess Body Weight and Outcome and Process Measures in Mechanically Ventilated Medical Intensive Care Unit Patients
Brief Title: Effects of Obesity on Care and Outcomes in Mechanically Ventilated Individuals in the Intensive Care Unit
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Ohio State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1330; K23HL075076 (NIH); K23HL075076-01A2 (NIH)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Respiratory Insufficiency
Keywords: Mechanical Ventilation; Critical Care; Respiratory Failure
MeSH Terms: conditions — Obesity; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Obesity is a significant health care issue in the United States, particularly among the critically ill. Preliminary research has shown that differences in ventilator management exist among obese and non-obese individuals. This study will examine the effect of excess weight on ventilator management and clinical outcomes in individuals in an intensive care unit (ICU).

DETAILED DESCRIPTION:
Sixty-four percent of American adults are overweight or obese. Excess weight will soon surpass smoking as the most common cause of preventable death. Despite the well-known health consequences of obesity, little is known about the specific effects of obesity in critically ill individuals. There are significant differences in ventilator management procedures among obese and non-obese individuals in an ICU. The long-term effect of these differences, however, has not been studied. Preliminary research has shown that differences in the mechanical ventilation process may be responsible for worse outcomes in obese individuals, as compared to non-obese individuals. The purpose of this study is to examine the effect of obesity on ventilator management processes and medical outcomes in individuals in an ICU. The study will also identify any increased risks for the critically ill obese and the causes of their augmented mortality and morbidity levels.

This study will enroll individuals in an ICU who are receiving mechanical ventilation through an endotracheal tube. Because potential participants are critically ill, and are unable to provide consent to participate in the study, each participant must have a surrogate decision maker who will provide consent on their behalf. Once enrolled, participants' weight, height, and waist circumference will be measured. Medical outcomes and information on the processes of ventilator management and care will be assessed while participants are in the ICU. Information on hospital outcomes, quality of life, utility, employment, and living situation will be collected upon release from the ICU, as well as during follow-up telephone interviews, which will occur every 90 days for a period of up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the ICU at Ohio State University Medical Center (OSUMC)
* Receiving mechanical ventilation through an endotracheal tube

Exclusion Criteria:

* Previously enrolled in this study
* Transferred from another acute care hospital
* Transferred from another ICU at OSUMC more than 24 hours after admission to that ICU
* Prisoner
* Unable to identify a surrogate decision maker or there is a dispute over who is the surrogate decision maker
* Pregnant
* Dies prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring mechanical ventilation admitted to the OSUMC MICU
Sampling Method: Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2006-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M. O'Brien, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] O'Brien JM Jr, Philips GS, Ali NA, Aberegg SK, Marsh CB, Lemeshow S. The association between body mass index, processes of care, and outcomes from mechanical ventilation: a prospective cohort study. Crit Care Med. 2012 May;40(5):1456-63. doi: 10.1097/CCM.0b013e31823e9a80. PMID 22430246